CLINICAL TRIAL: NCT02034734
Title: A Phase I, Open-label Study to Investigate the Safety, Tolerability and Plasma and Cerebrospinal Fluid Pharmacokinetics and Pharmacodynamics of Multiple Doses of ASP3652 in Healthy Young Caucasian Male Subjects
Brief Title: A Study to Investigate the Appearance and Disappearance of ASP3652 in Blood and Spinal Fluid in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3652-CL-0048; 2011-004226-97 (EudraCT Number)
Record Dates: First submitted 2014-01-10; First posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Pharmacokinetics of ASP3652; Pharmacodynamics of ASP3652; Healthy Subjects
Keywords: Phase 1; ASP3652; Cerebrospinal fluid (CSF); Multiple doses
MeSH Terms: interventions — ASP3652

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1: ASP3652 (Experimental): Multiple doses of ASP3652
  Interventions: Drug: ASP3652

INTERVENTIONS:
Drug: ASP3652 — oral

SUMMARY:
The purpose of this study is to evaluate the plasma and cerebrospinal fluid (CSF) pharmacokinetics (PK) of multiple doses of ASP3652 in healthy young Caucasian male subjects. Also to evaluate the plasma and CSF pharmacodynamics (PD) of multiple doses of ASP3652 in healthy young Caucasian male subjects and to assess the safety and tolerability of multiple doses of ASP3652 in healthy young Caucasian male subjects.

DETAILED DESCRIPTION:
Screening takes place between Day -22 to Day -2. Subjects are admitted to the clinical on Day -1 and remain until Day 12.

On Days 5 to 9, subjects receive twice-daily doses of ASP3652, and a single dose on the morning of Day 10. Subjects fast for 10h before the morning dose on Days 5 to 9 and they are served the first standard meal 1h after the morning dose.

A spinal tap is used to collect cerebrospinal fluid (CSF) on Day 1 and Day 10. A plasma sample for PK sample is obtained before first dosing on Day 5. To confirm steady-state concentrations of ASP3652 in plasma, blood samples are obtained before the morning dose on Days 7, 9 and 10, and before the evening dose on Days 5, 7 and 9. On Day 10, a PK profile of ASP3652 in plasma is obtained for up to 48h after the morning dose and for up to 24h in CSF.

Profiles of several enzyme substrates in plasma and seminal fluid (exploratory) are obtained on Day 1 and Day 10 up to 24h in CSF and up to 48h in plasma, before the morning and evening dose on Days 5, 7 and 9 in plasma.

Vital signs, 12-lead electrocardiograms (ECGs), safety laboratory assessments, adverse events (AEs) and concomitant medication are monitored throughout the investigational period until the ESV.

ELIGIBILITY:
Inclusion Criteria:

* Subject is white and of Caucasian origin.
* Body Mass Index more than or equal to 18.5 and less than 30.0 kg/m2.
* Male subject must agree to practice an adequate contraceptive method with female sexual partners to prevent pregnancy.

Exclusion Criteria:

* Known or suspected hypersensitivity to ASP3652 or any components of the formulation used.
* History of excessive bleeding or bruising.
* Abnormalities of coagulation screen including platelet count, prothrombin time (PT) and activated partial thromboplastin time (aPTT).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of ASP3652 in plasma measured by area under the plasma concentration-time curve in the dosing interval (AUCtau) | Days 5, 7 and 9, and Days 10 - 12
PK of ASP3652 in plasma measured by maximum observed plasma concentration (Cmax) | Days 5, 7 and 9, and Days 10 - 12
PK parameter of ASP3652 in cerebrospinal fluid (CSF) measured by area under the plasma concentration-time curve in the dosing interval (AUCtau) | Days 10 -11
PK parameter of ASP3652 in cerebrospinal fluid (CSF) measured by maximum observed plasma concentration (Cmax) | Days 10 -11

SECONDARY OUTCOMES:
Additional PK of multiple doses of ASP3652 in plasma and cerebrospinal fluid (CSF) | Plasma: Days 5, 7 and 9, and Days 10 - 12 / CSF: Days 10 -11
  plasma concentration immediately before the next dose (Ctrough), time to attain Cmax (tmax), apparent terminal elimination half-life (t½), volume of terminal phase distribution at steady state (Vz/F), apparent clearance after oral administration at steady state (CL/F) and peak trough ratio (PTR)
Pharmacodynamics (PD) of multiple doses of ASP3652 in plasma and CSF | Plasma: Days 1-3 and Days 5-12 / CSF: Days 1-2 and Days 10-11
  response immediately prior to dosing (Rtrough), time of the maximum response (tmaxR), maximum response (Rmax), area under the response-time curve from 0 to 12h (AURC0-12h), percentage change in maximum response (Rmax%), percentage change in AURC from 0 to 12h (AUR0-12h%)
Safety and tolerability of multiple doses of ASP3652 | Screening (Day -22 to Day -2) to End-of-Study Visit (7 to 14 days after (early) discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- PAREXEL Early Phase Clinical Unit, Harrow, United Kingdom

REFERENCES:
- [Derived] Takizawa M, Cerneus D, Michon I, Rijnders S, Meijer J, Someya A, Sato Y. Investigation of Safety and Tolerability of ASP3652 Based on Clinical Studies of Cerebrospinal Fluid Transfer After Multiple Doses and Exposure After Single Doses at High Dose Levels. Adv Ther. 2020 Sep;37(9):3967-3984. doi: 10.1007/s12325-020-01451-6. Epub 2020 Jul 26. PMID 32715381